CLINICAL TRIAL: NCT01662830
Title: Use of the Medifast Meal Replacement Program for Weight Loss in Obese Patients: A Restrospective Chart Review of Three Medifast Weight Control Centers (MWCC)
Brief Title: A Retrospective Chart Review of Three Medifast Weight Control Centers
Status: Completed | Type: Observational
Sponsor: Medifast, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MED 016
Record Dates: First submitted 2012-08-03; First posted 2012-08-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Obesity
Keywords: Obesity; Meal replacements
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MWCC clients: This study will be a systematic retrospective chart review of clients participating in the Jump Start (5 & 1) Plan at three different MWCC locations in Texas during the years 2007 - 2010.

SUMMARY:
The primary aim of this study is to to retrospectively evaluate the efficacy of the MWCC Jump Start (Medifast's 5 & 1) Plan on the following indices: weight loss, anthropometric changes, and reduction in common markers of coronary heart disease.

DETAILED DESCRIPTION:
Portion-controlled meal replacements by themselves have been shown to be an effective weight control strategy in overweight and obese individuals. The addition of medical supervision has been shown to result in greater weight loss than meal replacements alone. MWCC provides this added support through individual weekly counseling sessions. Thus, the investigators plan to retrospectively evaluate the efficacy of the MWCC Jump Start (Medifast's 5 & 1) Plan on the following indices: weight loss, anthropometric changes, and reduction in common markers of coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 18-70
* Followed the Jump Start (5 & 1) Plan
* BMI ≥ 25
* Purchased a weight management program at the MWCC location in the last 3 years
* Signed patient health information consent form

Exclusion Criteria:

* On a plan other than the 5&1 (Jump Start)
* Completed initial consultation but did not participate further
* Program stopped due to client not getting baseline labs
* Program stopped due for medical reasons unrelated to the 5 & 1 (Jump Start) plan
* Currently an active participant at the MWCC
* No signed patient health information consent form or written request to revoke consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study was a systematic retrospective chart review of patients participating in the Jump Start (5 & 1) Plan at three different MWCC locations in Texas during the years 2007-2010.
Sampling Method: Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Changes in weight | weeks 4, 12, 24 and final weight loss visit (average of 19.6 weeks)
  Weight loss (in pounds and percent weight loss) at weeks 4, 12, 24 and at final weight loss visit (average of 19.6 weeks).
Changes in body composition | weeks 4, 12, 24 and final weight loss visit (average of 19.6 weeks)
  changes in lean muscle mass, body fat mass, and body fat percent at weeks 4, 12, 24, and final weight loss visit(average of 19.6 weeks).

SECONDARY OUTCOMES:
Compliance | weeks 4, 12, 24 and final weight loss visit (average of 19.6 weeks)
  Compliance is measured by client attendance at weekly visits, consumption of meal replacements and dietary supplements, ketone testing, and completion of food journals
Retention rates | weeks 4, 12, 24 and final weight loss visit (average of 19.6 weeks)
  Retention of clients at specified time points (weeks 4, 12, 24 and final weight loss visit) and during the transition and weight maintenance phases of the MWCC weight management program
Goal weight achievement | Final weight loss visit (average of 19.6 weeks)
  The percent of clients that achieve thier goal weight by their final weight loss visit(average of 19.6 weeks)
Changes in abdominal circumference (inches) | weeks 4, 12, 24 and final weight loss visit (average of 19.6 weeks)
Maintenance of weight loss | Following transition (up to 12 weeks) and maintenance (up to 52 weeks) phases of the program
Changes in cardiovascular risk factors | weeks 4, 12, 24 and final weight loss visit (average of 19.6 weeks)
  Improvements in diastolic and systolic blood pressure and pulse at weeks 4, 12, 24 and final weight loss visit (average of 19.6 weeks).

REFERENCES:
- [Background] Heymsfield SB, van Mierlo CA, van der Knaap HC, Heo M, Frier HI. Weight management using a meal replacement strategy: meta and pooling analysis from six studies. Int J Obes Relat Metab Disord. 2003 May;27(5):537-49. doi: 10.1038/sj.ijo.0802258. PMID 12704397
- [Background] Haddock CK, Poston WS, Foreyt JP, DiBartolomeo JJ, Warner PO. Effectiveness of Medifast supplements combined with obesity pharmacotherapy: a clinical program evaluation. Eat Weight Disord. 2008 Jun;13(2):95-101. doi: 10.1007/BF03327609. PMID 18612258